CLINICAL TRIAL: NCT03140982
Title: Is Anesthetic Loss of Consciousness a Cortical or Brainstem Phenomenon? What Does the Neurological Examination Say?
Brief Title: Is Anesthetic Loss of Consciousness a Top Down or Bottom up Phenomenon. What Does the Neurologic Examination Say?.
Acronym: Top&Bottom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Pablo O. Sepulveda, MD. Professor in Anesthesia, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Centro Bioetica 2016-05
Record Dates: First submitted 2017-04-10; First posted 2017-05-04 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia; Functional
Keywords: propofol; pharmacology; anesthesic induction; drug titration
MeSH Terms: interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: comparison of the neurologic behavior between two group, a fast and a slow anesthesia induction
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: after patient constent, and previos the patient arriving the OR, the care provider (designed anesthestist) using a coin decide the arm (GR or GL). The neurologist and investigator was blind to the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GR fast induction (Active Comparator): propofol TCI effect site mode infusion using the PK Marsh model ke0 1,21 min-1 target 5.4 ug/ml (LOC EC95) util loss of consciousness (LOC) After LOC we maintain initial target during 10 min without intervention, except respiratory support if required.
  Interventions: Diagnostic Test: FOUR coma scale and frontal espectrograpy evaluation
- GL slow induction (Active Comparator): propofol infused at 10 mg/kg/h with CeCALC PK Marsh model ke0 1,21 min-1 same PK model After LOC we maintain the CeCALC observed al LOC during 10 min without intervention, except respiratory support if it was required.
  Interventions: Diagnostic Test: FOUR coma scale and frontal espectrograpy evaluation

INTERVENTIONS:
Diagnostic Test: FOUR coma scale and frontal espectrograpy evaluation — systematic evaluation using the validated FOUR coma scale during propofol administration
  Other Names: 4 channel EEG record with SEDline monitor; Non Invasive Blood presure, Saturation 02, Electrocardiogram; propofol infusion in Target controlled infusion using Primea Orchestra infusion pump Fressenius Kabi

SUMMARY:
Using very slow or fast propofol intravenous injection, monitored using standard American Society of Anesthesiology (ASA) standard and SEDLine EEG (Med Tech), the patient was evaluate by a neurologist every 30 sec using the FOUR coma scale.

DETAILED DESCRIPTION:
Clinical experimental randomized study, approved by the Ethic Committee, with informed consent, included ASA I- II adults, without neurological illness and normal physical exam.

The patient randomized in two groups, rapid induction (GR) with propofol in target controlled infusion (TCI) effect site mode using the phamacokinetic (PK) model from Marsh ke0 1,21 min-1 using a calculated target of 5.4 ug/ml (loss of counsciousness EC95) and slow induction (GL) 10 mg/kg/h with calculated effect site concentrations (CeCALC) same PK model.

The same neurologist, blind to the correspondent group, evaluated all the patients every 30 sec using the coma FOUR scale until loss of counsciousness (LOC), defined as a FOUR (E0 no eyes opening response and /or M0 no motor response). At LOC the existance of brainstem reflex was evaluated (B no pupil and corneal reflex), respiratory pattern (R apnoea), CeCALC and patient state index (PSI) SEDline™ was recorded during all the examination.

After LOC in both groups we maintain in GR the initial target (5.3 ug/ml) and the LOC CeCALC during 10 min without intervention, except respiratory support if it was required.

Frontal EEG 4 channel and spectrogram from SEDline monitor was extracted for each case and posterior analysis.

Fisher exact test was used to describe primary outcome and difference between B and R for each group. The difference in time to reach LOC LOC, Ce and PSI was analysed with T- Student.

ELIGIBILITY:
Inclusion Criteria: ASA 1-2 patients programmed for elective surgery, normal neurologic examination -

Exclusion Criteria: neurologic illness, receiving drugs that affect Central Nervous System during the last 48 hours

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
loss of consciousness a cortical or brainsteam phenomenon | 1 year
  with fast and slow induction we use the FOUR coma scale ( Ann Neurol. 2005;58(4): 585-93) to identify lost of brain stem activities.

SECONDARY OUTCOMES:
evaluation of the alfa band behavior after fast and slow inductions | 1 year
  the investigators analyze the time delay in stabilizing the frontal alfa band after fast and slow anesthesia inductions

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lavados, MD, Study Chair — Clinica Alemana Comité Cientifico
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Mashour GA. Top-down mechanisms of anesthetic-induced unconsciousness. Front Syst Neurosci. 2014 Jun 23;8:115. doi: 10.3389/fnsys.2014.00115. eCollection 2014. PMID 25002838
- [Background] Wijdicks EF, Bamlet WR, Maramattom BV, Manno EM, McClelland RL. Validation of a new coma scale: The FOUR score. Ann Neurol. 2005 Oct;58(4):585-93. doi: 10.1002/ana.20611. PMID 16178024